CLINICAL TRIAL: NCT03321032
Title: Second-generation drUg-elutinG Stents in diAbetes: a Randomized Trial (the SUGAR Trial)
Brief Title: Second-generation Drug-eluting Stents in Diabetes
Acronym: SUGAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Dr Rafael Romaguera, Principal Investigator, Spanish Society of Cardiology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEC-SUG-2016-01
Record Dates: First submitted 2017-10-22; First posted 2017-10-25 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: Coronary Artery Disease; Diabetes Mellitus; Drug-eluting stents; Restenosis
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amphilimus-eluting stents (Experimental): Polymer-free Amphilimus-eluting stents
  Interventions: Device: Polymer-free amphilimus-eluting stents
- Zotarolimus-eluting stents (Active Comparator): Biolinx Polymer-based zotarolimus-eluting stents
  Interventions: Device: Biolinx Polymer-based zotarolimus-eluting stents

INTERVENTIONS:
Device: Polymer-free amphilimus-eluting stents — Cre8 Evo coronary stent system (CID, Saluggia, Italy)
  Arms: Amphilimus-eluting stents
Device: Biolinx Polymer-based zotarolimus-eluting stents — Resolute Onyx coronary stent system (Medtronic, Minneapolis, Minnesota, US)
  Arms: Zotarolimus-eluting stents

SUMMARY:
This is an investigator initiated randomized trial, performed under the auspices of the Spanish Society of Cardiology.

It is a multicenter, international, parallel, randomized 1:1 (amphilimus-eluting stents vs zotarolimus-eluting stents) clinical trial performed exclusively in patients with diabetes mellitus. The study has an "all-comers diabetics" design.

The primary-endpoint is target lesion failure at 1-year follow-up (non-inferiority design) and the co-primary end-point is target lesion failure at 2-years follow-up (superiority-design).

ELIGIBILITY:
Inclusion Criteria(must meet all):

* Patients ≥18 years who understands the nature of the study and provides written informed consent.
* Diagnosis of diabetes according to the American Diabetes Association diagnostic criteria (*)
* Documented silent ischemia, stable angina, unstable angina, or myocardial infarction (with or without ST elevation).
* At least one de novo coronary lesion with stenosis of more than 50% in a vessel with a reference vessel diameter of 2.25 to 4.5 mm by visual estimation. Coronary anatomy is suitable for PCI (patients with potential CABG indication should be eligible for PCI after a multidisciplinary evaluation in a Heart Team).

Exclusion Criteria:

* Cardiogenic shock or resuscitation
* Comorbidity with anticipated life expectancy to 24 months
* Inability to consent due to mechanical ventilation
* Pregnant female patient
* Conditions that could preclude a minimal of 1 month of DAPT (such as, but not limited to: severe liver failure, platelet count <100,000 cells/mm3, recent gastrointestinal bleeding or history of bleeding diathesis or coagulopathy)
* Contraindication or known allergy to aspirin, heparin, P2Y12 inhibitors, cobalt and/or chromium metal alloys, sirolimus or derivates, polyurethane, or contrast media (for contrast-media allergy, patients that might be safely and adequately pre-medicated should be allowed to enter the study).
* Currently enrolled in another clinical trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2021-01-28 (Estimated); Study Completion 2022-01-28 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure at 1-year follow-up | 12 months
  A composite of cardiac death, any myocardial infarction (not clearly attributable to a non-target vessel), or clinically indicated target-lesion revascularization at 12-months follow-up.
Target lesion failure at 2-years follow-up | 24 months
  A composite of cardiac death, any myocardial infarction (not clearly attributable to a non-target vessel), or clinically indicated target-lesion revascularization at 24-months follow-up.

SECONDARY OUTCOMES:
Cardiac death | 12 and 24 months
Target vessel myocardial infarction | 12 and 24 months
Target vessel revascularization | 12 and 24 months
Target lesion revascularization | 12 and 24 months
Stent thrombosis | 12 and 24 months
  Academic Research Consortium definitions
Non-target lesion revascularization | 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (23):
- Spain (23):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital San Juan, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Doctor Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario de León, León
  - Hospital Lucus Augusti, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Clínica Universidad de Navarra, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Marqués de Valdecilla, Santander
  - Hospital de Santiago, Santiago de Compostela
  - Hospital Joan XXIII, Tarragona
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico de Valencia, Valencia
  - Hospital Álvaro Cunqueiro, Vigo

REFERENCES:
- [Result] Romaguera R, Salinas P, Brugaletta S, Gomez-Lara J, Diaz JF, Romero MA, Garcia-Blas S, Ocaranza R, Borde P, Jimenez Kockar M, Millan Segovia R, Iniguez A, Alameda M, Trillo R, Lee DH, Martin P, Lopez-Benito M, Frutos A, Moreu J, Hernandez-Hernandez F, Garcia Del Blanco B, Roura G, Rossello X, Pocock SJ, Fernandez-Ortiz A, Sabate M, Gomez-Hospital JA. Second-Generation Drug-Eluting Stents in Diabetes (SUGAR) trial: Rationale and study design. Am Heart J. 2020 Apr;222:174-182. doi: 10.1016/j.ahj.2020.01.018. Epub 2020 Jan 28. No abstract available. PMID 32087418
- [Derived] Salinas P, Romaguera R, Gomez-Lara J, Brugaletta S, Gomez-Menchero A, Martin P, Romero M, Garcia-Blas S, Jimenez M, Jimenez VA, Bordes P, Bayon J, Salvatella N, Alameda M, Hyun-Lee D, Trillo-Nouche R, Lopez-Benito M, Frutos A, Moreu J, Garcia Del Blanco B, Mohandes M, Bosa Ojeda F, Hernandez Hernandez F, Pinar-Bermudez E, Jimenez-Quevedo P, Rossello X, Pocock S, Sabate M, Gomez-Hospital JA, Comin-Colet J, Gonzalo N, Fernandez Ortiz A; SUGAR trial Investigators. Amphilimus-eluting versus zotarolimus-eluting stents in patients with diabetes mellitus and coronary artery disease: extended follow-up of the SUGAR randomised controlled trial. Heart. 2025 Nov 25;111(24):1191-1198. doi: 10.1136/heartjnl-2025-325773. PMID 40562528
- [Derived] Romaguera R, Salinas P, Gomez-Lara J, Brugaletta S, Gomez-Menchero A, Romero MA, Garcia-Blas S, Ocaranza R, Bordes P, Kockar MJ, Salvatella N, Jimenez-Diaz VA, Alameda M, Trillo R, Lee DH, Martin P, Lopez-Benito M, Freites A, Pascual-Tejerina V, Hernandez-Hernandez F, Blanco BGD, Mohandes M, Bosa F, Pinar E, Roura G, Comin-Colet J, Fernandez-Ortiz A, Macaya C, Rossello X, Sabate M, Pocock SJ, Gomez-Hospital JA; SUGAR trial investigators. Amphilimus- vs. zotarolimus-eluting stents in patients with diabetes mellitus and coronary artery disease: the SUGAR trial. Eur Heart J. 2022 Mar 31;43(13):1320-1330. doi: 10.1093/eurheartj/ehab790. PMID 34735004